CLINICAL TRIAL: NCT04964544
Title: A Phase III, 6-Month Self-selection and Actual Use Study for Rx-to-OTC Switch of Rosuvastatin 5 mg Once-daily in Combination With a Web App
Brief Title: Technology-Assisted Cholesterol Trial in Consumers (TACTiC)
Acronym: TACTiC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Concentrics Research (Other); Idea Evolver (Industry); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D356PL00015
Record Dates: First submitted 2021-06-22; First posted 2021-07-16 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: High Cholesterol
Keywords: Cholesterol, Web App
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: This is a 6-month, single-arm, uncontrolled technology-assisted Self-Selection and Actual Use Study to evaluate the use of nonprescription rosuvastatin 5 mg in combination with a Web App. It is an open-label study where participants qualify for treatment based on the medical history, laboratory and blood pressure data they enter into the Web App, accessed on their own device on the internet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label, Single Arm Technology-Assisted Cholesterol Trial (Other): Open Label Single Arm study in All-comers population who self-report having concern about high cholesterol or heart health
  Interventions: Combination Product: 5 mg rosuvastatin calcium with a Web App (combination product)

INTERVENTIONS:
Combination Product: 5 mg rosuvastatin calcium with a Web App (combination product) — The combination product will be a Drug (Rosuvastatin calcium 5 mg) and Software as a Medical Device (Web App that features a Technology-Assisted Self-Selection (TASS) tool). Rosuvastatin calcium 5 mg will be taken orally, 1 tablet daily to use for lowering cholesterol, a key risk factor that can lead to heart disease.
  Other Names: Crestor 5 mg

SUMMARY:
The purpose of this AUS is to evaluate the extent to which participants can safely and effectively self-select, purchase, and use Crestor OTC 5 mg for a 6-month period according to the label.

DETAILED DESCRIPTION:
This is a single-arm, interventional, phase III Self-Selection (SS) and Actual Use Study (AUS) using a technology assisted tool within a Web App. The open-label study will enroll approximately 1220 participants who qualify for treatment based on the data they enter into the Web App of which an estimated 1000 participants will ultimately proceed to the use phase.

ELIGIBILITY:
Inclusion Criteria:

1. Males, 20-75 years of age
2. Females, 20-75 years of age (This inclusion criterion will be applied until 50 females under the age of 50 years complete the initial TASS assessment in the Web App). After this quota of 50 females under the age of 50 years old is met, the inclusion criterion will be revised to females 50-75 years old).
3. Respond to advertising regarding a concern about high cholesterol or heart health
4. Able to read speak and understand English

Additional Criteria for Inclusion for Actual Use (at Virtual Visit 1)

1. Participant reads and signs the Informed Consent form

Exclusion Criteria:

1. The participant or anyone in their household is currently employed by any of the following:

   * A pharmacy or pharmaceutical company
   * A consumer healthcare company
   * A manufacturer of medicines
   * A managed care or health insurance company
   * A healthcare practice
   * An employee of AstraZeneca or Concentrics Research
2. The participant has ever been trained or employed as a healthcare professional (physician, nurse, nurse practitioner, physician assistant, pharmacist).
3. The participant has, or cannot recall whether he/she has, received an investigational therapy as part of a clinical trial in the previous twelve (12) months
4. The participant is not willing to provide contact information.
5. Previous enrollment in the present study.
6. The participant has a mailing address in Alaska or their mailing address is a Post Office (PO) Box.
7. The participant is not willing to complete an eDiary
8. The participant is a woman of childbearing potential and is not following contraception guidelines or is not willing to follow contraception guidelines including practicing abstinence or using at least 1 of the following acceptable methods of birth control for at least 1 month prior to entry into the study and for 1 month after study completion: hormonal -oral, implantable, injectable, or transdermal; mechanical - spermicide in conjunction with a barrier such as a condom or diaphragm; intrauterine device; or surgical sterilization of partner.
9. The participant does not have access to the internet.
10. The participant does not have an email address or the ability to receive emails.
11. The participant responds to the Single Item Literacy Screener 2 (SILS2) question (See References) with either 'extremely' or 'quite a bit.' (If the quota for normal literacy is met, but the limited literacy target is not met, the SILS2 exclusion will be used to help increase the percentage of limited literacy participants at Virtual Visit 1. Participants identified as normal literacy by Rapid Estimate of Adult Literacy in Medicine [REALM] testing at Virtual Visit 1 will not be excluded from entry into the treatment phase of the study.)
12. Inability to conduct interviews in a private location so that sensitive information about the participant or study would not be overheard by others not permitted to hear such information.

Additional Criteria for Exclusion from Actual Use (at Virtual Visit 1)

Confirmation by Concentrics Central Medical Operations Group (CMOG) clinician:

1. That the participant is pregnant, as determined by an approved self-administered OTC urine pregnancy test (UPT) conducted for all female participants of childbearing potential (Female participants who are not post-menopausal or surgically sterile).
2. That the participant is breastfeeding.
3. That the participant has an allergy to rosuvastatin.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1196 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C. Miller, M.D., Principal Investigator — Concentrics Central Medical Operations Group
Locations (1):
- Research Site, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] Chew LD, Griffin JM, Partin MR, Noorbaloochi S, Grill JP, Snyder A, Bradley KA, Nugent SM, Baines AD, Vanryn M. Validation of screening questions for limited health literacy in a large VA outpatient population. J Gen Intern Med. 2008 May;23(5):561-6. doi: 10.1007/s11606-008-0520-5. Epub 2008 Mar 12. PMID 18335281
- [Background] Davis TC, Long SW, Jackson RH, Mayeaux EJ, George RB, Murphy PW, Crouch MA. Rapid estimate of adult literacy in medicine: a shortened screening instrument. Fam Med. 1993 Jun;25(6):391-5. PMID 8349060
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Jun 18;139(25):e1082-e1143. doi: 10.1161/CIR.0000000000000625. Epub 2018 Nov 10. PMID 30586774
- [Derived] Nissen SE, Hutchinson HG, Wolski K, Watson K, Martin SS, Michos ED, Weintraub WS, Morris M, Cho L, Laffin L, Jacoby D, Ballantyne CM, Ekelund J, Birve F, Menon V, Strzelecki M, Ridker PM. A Technology-Assisted Web Application for Consumer Access to a Nonprescription Statin Medication. J Am Coll Cardiol. 2024 May 28;83(21):2080-2088. doi: 10.1016/j.jacc.2024.03.388. Epub 2024 Apr 8. PMID 38599257
- See also: Study Landing Page — http://lowercholesterol.study
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D356PL00015&attachmentIdentifier=c0a32e33-61a7-46a8-9711-1dc23e122ebb&fileName=redacted_CSP.pdf&versionIdentifier=
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D356PL00015&attachmentIdentifier=a51da88d-0773-4001-b444-d89a9aab4c08&fileName=redacted_SAP.pdf&versionIdentifier=
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D356PL00015&attachmentIdentifier=bad1de2a-9917-447a-aabd-2dd5c5bf45e7&fileName=redacted_CSR_Synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Nonprescription Rosuvastatin: Combination Product: 5 mg rosuvastatin calcium with a Web App (combination product)
Period: Overall Study
Arm/Group | Nonprescription Rosuvastatin
Started | 1196
Had an Ask a Doctor Before Use Warning Identified by the CMOG at Final Use Visit | 25
Had a do Not Use Warning Identified by the CMOG at Final Use Visit | 59
Participants for Whom CMOG Identified a Stop Use Warning at Final Use Assessment | 2
Completed | 1154
Not Completed | 42
Not completed — Screen failure or other uncategorised | 10
Not completed — Physician Decision | 4
Not completed — Lost to Follow-up | 9
Not completed — Withdrawal by Subject | 18
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nonprescription Rosuvastatin
Number analyzed (Participants) | 1196
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The full analysis set population
  Years | 61.6 (8.1)
Age, Customized [Count of Participants; unit: Participants]
  Under 20 years of age | 0
  20-29 years of age | 4
  30-39 years of age | 18
  40-49 years of age | 64
  50-59 years of age | 334
  60-69 years of age | 598
  70-75 years of age | 178
  76+ years of age | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The full analysis set population
  Participants
    Female | 474
    Male | 722
Race/Ethnicity, Customized [Number; unit: Participants] — Population: The full analysis set population
  Participants
    White | 949
    Hispanic | 38
    Black or African American | 140
    Asian (China, Philippines, Vietnam, Korea, etc.) | 34
    South Asian (India, Pakistan, Bangladesh, etc.) | 14
    Other | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Correct Initial TASS Outcome, Worst Case Imputation, First Co-Primary Endpoint (Self-Selection Population)
Description: Proportion of participants that had a correct tass outcome at their initial TASS assessment
Time Frame: Study day -30 to -1, at initial TASS assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Nonprescription Rosuvastatin
Number analyzed (Participants) | 1196
Participants | 1085
Statistical Analysis 1: Comparison: Nonprescription Rosuvastatin; Proportion of participants with overall correct initial TASS assessment, with mitigations, worst case imputation (Self-Selection Population); Test type: Other; Percentage = 90.7, 95% CI 2-sided [88.9 to 92.3] — Proportion of participants

2. Primary Outcome: Overall Correct Final Use Outcome With Mitigation, Second Co-primary Endpoint (Per Protocol Population)
Description: Proportion of participants that had a correct tass outcome at their final TASS assessment
Time Frame: From enrollment to end of the home use period at 180 days, at final TASS Assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Nonprescription Rosuvastatin
Number analyzed (Participants) | 1154
Participants | 1132
Statistical Analysis 1: Comparison: Nonprescription Rosuvastatin; Proportion of participants with overall correct final TASS assessment, with mitigations, worst case imputation (Per Protocol Population); Test type: Other; Percentage = 98.1, 95% CI 2-sided [97.1 to 98.8] — Proportion of participants

3. Primary Outcome: Percent Change From Baseline in Verified LDL-C Regardless of Final Use Outcome (AUS ITT Population)
Time Frame: From enrollment to end of the home use period at 180 days, at final assessment
Measure: Mean (95% Confidence Interval); unit: Percent change of baseline
Arm/Group | Nonprescription Rosuvastatin
Number analyzed (Participants) | 1063
Percent change of baseline | -35.48 [-36.63 to -34.33]
Statistical Analysis 1: Comparison: Nonprescription Rosuvastatin; Test type: Other; Mean percent change from paseline = -35.48, 95% CI 2-sided [-36.63 to -34.33]

4. Secondary Outcome: Participants Eligble for Continuous Treatment Who Self-Tested With a Verified LDL-C Retest During Study, Overall and by Subgroups (Per Protocol Population)
Time Frame: From enrollment to end of the home use period at 180 days
Population: Participants in the per protocol analysis set eligble for continuous treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nonprescription Rosuvastatin
Number analyzed (Participants) | 910
Participants | 845

5. Secondary Outcome: Participants Who Self-Identify a Stop Use Warning Also Identified by the CMOG, and Stop Medication (Per Protocol Population)
Description: Participants who Self-Identify a Stop Use Warning also identified by the CMOG, and Stop Medication.
Time Frame: From enrollment to end of the home use period at 180 days
Population: Participants who had a stop use warning identified by the CMOG at final use assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Nonprescription Rosuvastatin
Number analyzed (Participants) | 2
Participants | 1

6. Secondary Outcome: Participants Who Self-Identify a Do Not Use Warning Also Identified by the CMOG at Final Use Assessment(Per Protocol Population, Participants Who Had a do Not Use Warning Identified by the CMOG at Final Use Visit)
Time Frame: From enrollment to end of the home use period at 180 days
Population: Participants in the per protocol population who had a do not use warning identified by the CMOG at final use visit
Measure: Count of Participants; unit: Participants
Arm/Group | Nonprescription Rosuvastatin
Number analyzed (Participants) | 59
Participants | 46

7. Secondary Outcome: Participants Who Self-Identify an Ask a Doctor Before Use Warning Also Identified by the CMOG at Final Use Assessment (Per Protocol Population, Participants Who Had a do Not Use Warning Identified by the CMOG at Final Use Visit)
Time Frame: From enrollment to end of the home use period at 180 days
Population: Participants in the per protocol population who had an ask a doctor before use warning identified by the CMOG at final use visit
Measure: Count of Participants; unit: Participants
Arm/Group | Nonprescription Rosuvastatin
Number analyzed (Participants) | 25
Participants | 23

8. Secondary Outcome: Participants With Overall Compliance Between 50% and 120%
Description: Overall compliance is defined as 100 * (total number of pills taken) / (Intended duration of treatment in days)
Time Frame: From enrollment to end of the home use period at 180 days
Population: Participants in the per protocol population whose overall compliance was assessed
Measure: Count of Participants; unit: Participants
Arm/Group | Nonprescription Rosuvastatin
Number analyzed (Participants) | 1146
Participants | 1089

9. Secondary Outcome: Participants Who Were Longitudinally Compliant (Per Protocol Population)
Description: An individual is longitudinally compliant if they have 50% to 120% compliance across each supply period.
Time Frame: From enrollment to end of the home use period at 180 days
Population: Participants in the per protocol population for whom supply period compliance was assessed across all supply periods
Measure: Count of Participants; unit: Participants
Arm/Group | Nonprescription Rosuvastatin
Number analyzed (Participants) | 1134
Participants | 848

10. Secondary Outcome: Participants Who Were Persistent (Per Protocol Population)
Description: An individual is persistent if they ordered the full 180 days of treatment and were eligible for continuous treatment
Time Frame: From enrollment to end of the home use period at 180 days
Population: Participants in the per protocol population that were eligible for continuous treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nonprescription Rosuvastatin
Number analyzed (Participants) | 910
Participants | 896

ADVERSE EVENTS:
Time Frame: treatment period (6 months)
Arm/Group | Nonprescription Rosuvastatin
All-Cause Mortality (participants affected / at risk) | 1/1177
Serious Adverse Events (participants affected / at risk) | 27/1177
Other Adverse Events (participants affected / at risk) | 493/1177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nonprescription Rosuvastatin (N=1177)
Gastric ulcer (Gastrointestinal disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chromophobe renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Aortic aneurysm (Vascular disorders) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nonprescription Rosuvastatin (N=1177)
Nausea (Gastrointestinal disorders) | 26 (27)
Fatigue (General disorders) | 49 (52)
Pain (General disorders) | 32 (33)
Pyrexia (General disorders) | 21 (21)
Covid-19 (Infections and infestations) | 17 (17)
Sinusitis (Infections and infestations) | 13 (13)
Suspected covid-19 (Infections and infestations) | 14 (14)
Urinary tract infection (Infections and infestations) | 26 (27)
Sars-cov-2 test positive (Investigations) | 126 (129)
Arthralgia (Musculoskeletal and connective tissue disorders) | 83 (113)
Back pain (Musculoskeletal and connective tissue disorders) | 41 (44)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 41 (51)
Myalgia (Musculoskeletal and connective tissue disorders) | 49 (66)
Neck pain (Musculoskeletal and connective tissue disorders) | 14 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 51 (59)
Dizziness (Nervous system disorders) | 22 (22)
Headache (Nervous system disorders) | 69 (81)
Cough (Respiratory, thoracic and mediastinal disorders) | 50 (52)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 15 (17)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 28 (30)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 30 (33)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Rash (Skin and subcutaneous tissue disorders) | 14 (14)
Hypertensive urgency (Vascular disorders) | 20 (20)
Constipation (Gastrointestinal disorders) | 17 (18)
Diarrhoea (Gastrointestinal disorders) | 41 (47)

LIMITATIONS AND CAVEATS:
TACTiC was conducted during the COVID-19 pandemic. However, the pandemic was not judged to adversely impact the quality of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings. If this is foreseen, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT04964544/Prot_002.pdf
  • Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT04964544/SAP_001.pdf